CLINICAL TRIAL: NCT01881230
Title: A Phase 2/3, Multi-Center, Open-Label, Randomized Study of Weekly Nab®-Paclitaxel in Combination With Gemcitabine or Carboplatin, Compared to Gemcitabine/Carboplatin, as First Line Treatment in Subjects With ER, PgR, and HER2 Negative (Triple Negative) Metastatic Breast Cancer
Brief Title: Evaluate Risk/Benefit of Nab Paclitaxel in Combination With Gemcitabine and Carboplatin Compared to Gemcitabine and Carboplatin in Triple Negative Metastatic Breast Cancer (or Metastatic Triple Negative Breast Cancer)
Acronym: tnAcity
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABI-007-MBC-001; 2013-000113-20 (EudraCT Number)
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Results first posted 2018-03-08 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Breast Tumor; Breast Cancer; Cancer of the Breast; Estrogen Receptor- Negative Breast Cancer; HER2- Negative Breast Cancer; Progesterone Receptor- Negative Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer; Triple-negative Breast Cancer; Triple-negative Metastatic Breast Cancer; Metastatic Breast Cancer
Keywords: Breast Cancer; Cancer of the Breast; Metastatic Breast Cancer; Metastatic Triple Negative Breast Cancer; Triple Negative Breast Cancer; Triple Negative Metastatic Breast Cancer; Basal-like breast cancer; Hormone receptor negative breast cancer; Estrogen receptor negative breast cancer; Progesterone negative receptor breast cancer; HER2 Negative Breast Cancer; Abraxane; nab-Paclitaxel; ABI-007; gemcitabine; Gemzar; carboplatin; Paraplatin; Paraplatin AQ; Phase 2; Phase 3
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- nab-Paclitaxel plus Gemcitabine (Experimental): Treatment Arm A: nab-Paclitaxel 125 mg/m^2 by intravenous (IV) administration over 30 minutes, followed by gemcitabine 1000 mg/m^2 on Days 1 and 8 of each 21-day cycle by IV administration over 30 minutes
  Interventions: Drug: nab-Paclitaxel; Drug: Gemcitabine
- nab-Paclitaxel plus Carboplatin (Experimental): Treatment Arm B: nab-Paclitaxel 125 mg/m^2 on Days 1 and 8 by IV administration followed by carboplatin at an Area Under the Curve (AUC) of 2 on Days 1 and 8 of each 21-day cycle by IV administration
  Interventions: Drug: nab-Paclitaxel; Drug: Carboplatin
- Gemcitabine plus Carboplatin (Active Comparator): Treatment Arm C: Gemcitabine 1000 mg/m^2 on Days 1 and 8 by IV administration followed by carboplatin AUC 2 on Days 1 and 8 of each 21-day cycle by IV administration
  Interventions: Drug: Carboplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: nab-Paclitaxel — nab-Paclitaxel 125 mg/m^2 by IV administration over 30 minutes on Days 1 and 8 of each 21-day treatment cycle.
  Other Names: Abraxane
  Arms: nab-Paclitaxel plus Carboplatin; nab-Paclitaxel plus Gemcitabine
Drug: Carboplatin — Carboplatin at an AUC of 2 on Days 1 and 8 of each 21-day cycle by IV administration
  Other Names: Paraplatin,; Paraplatin AQ
  Arms: Gemcitabine plus Carboplatin; nab-Paclitaxel plus Carboplatin
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 on Days 1 and 8 of each 21-day treatment cycle.
  Other Names: Gemzar
  Arms: Gemcitabine plus Carboplatin; nab-Paclitaxel plus Gemcitabine

SUMMARY:
The purpose of this study is to compare the safety and efficacy of nab-paclitaxel in combination with either gemcitabine or carboplatin to the combination of gemcitabine and carboplatin as first line treatment in female subjects with triple negative metastatic breast cancer (TNMBC) or metastatic triple negative breast cancer.

DETAILED DESCRIPTION:
ABI-007-MBC- 001 is a Phase 2/3, multicenter, open-label, randomized, study that will compare the safety and efficacy of weekly nab-paclitaxel in combination with gemcitabine or carboplatin to the combination of gemcitabine and carboplatin as first line therapy in female subjects with Estrogen Receptor (ER), Progesterone Receptor (PgR), and human epidermal growth factor receptor 2 (HER2) negative (triple negative) metastatic breast cancer (TNMBC) or metastatic triple negative breast cancer. In the phase 2 portion of the study, the combinations of nab-paclitaxel plus gemcitabine and nab-paclitaxel plus carboplatin will be evaluated, and a comparator arm of gemcitabine combined with carboplatin will be used. In the phase 3 portion of the study, the selected nab-paclitaxel combination treatment will be compared to gemcitabine combined with carboplatin to evaluate progression free survival, safety and tolerability, overall survival, disease control rate and duration of response in women with metastatic triple negative breast cancer.

Due to changes in the treatment landscape since the initiation of this trial, the decision was made not to proceed to the Phase 3 portion of the study.

ELIGIBILITY:
Inclusion Criteria: A subject will be eligible for inclusion in this study only if all of the following criteria are met:

1. Female subjects, age ≥ 18 years at the time informed consent is signed
2. Pathologically confirmed adenocarcinoma of the breast
3. Pathologically confirmed as triple negative, source documented, defined as both of the following

   1. Estrogen Receptor (ER) and Progesterone Receptor (PgR) negative: < 1% of tumor cell nuclei are immunoreactive in the presence of evidence that the sample can express ER or PgR (positive intrinsic controls)
   2. Human Epidermal Growth Factor Receptor 2 (HER2) negative as per American Society of Clinical Oncology - College of American Pathologists (ASCO/CAP) guidelines i. Immunohistochemistry (IHC) 0 or 1 Fluorescence In Situ Hybridization (FISH) negative (or equivalent negative test). Subjects with IHC 2 must have a negative by Fluorescence In Situ Hybridization (FISH),, (or equivalent negative test).
4. Subjects with prior breast cancer history of different phenotypes (ie, ER/PgR/HER2 positive) must have pathologic confirmation of triple negative disease in at least one of the current sites of metastasis
5. Subjects must have received prior adjuvant or neoadjuvant anthracycline therapy; unless (a) anthracycline treatment was not indicated or was not the best treatment option for the subject in the opinion of the treating physician; and (b) anthracycline treatment remains not indicated or, in the opinion of the treating physician, is not the best treatment option for the subject's metastatic disease.

   a. Newly diagnosed subjects presenting with TNMBC are eligible for the study if anthracycline treatment is not indicated or is not the best treatment option for the subject in the opinion of the treating physician.
6. Subjects with measurable metastatic disease, defined by Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) guidelines
7. Life expectancy ≥ 16 weeks from randomization
8. No prior cytotoxic chemotherapy for metastatic breast cancer. Prior immunotherapy and/or monoclonal antibody therapy are acceptable. Prior treatments must have been discontinued at least 30 days prior to start of study treatment and all related toxicities must have resolved to Grade 1 or less.
9. Prior neoadjuvant or adjuvant chemotherapy, if given, must have been completed at least 6 months before randomization with all related toxicities resolved, and documented evidence of disease progression per RECIST 1.1 guidelines is required.

   a. If prior neoadjuvant or adjuvant chemotherapy contained taxane, gemcitabine, or platinum agents, the treatment must have completed at least 12 months before randomization
10. Prior radiotherapy must have completed before randomization, with full recovery from acute radiation side effects. At least one measurable lesion must be completely outside the radiation portal or there must be unequivocal radiologic or clinical exam proof of progressive disease within the radiation portal, in accordance with RECIST 1.1 guidelines
11. At least 30 days from major surgery before randomization, with full recovery
12. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
13. Subject has the following blood counts at screening:

    * Absolute Neutrophil Count (ANC) ≥ 1500/mm^2 ;
    * Platelets ≥ 100,000/mm^2 ;
    * Hemoglobin (Hgb) ≥ 9 g/dL
14. Subject has the following blood chemistry levels at screening:

    * Aspartate aminotransferase (AST) Serum glutamic-oxaloacetic transaminase (SGOT), Alanine Aminotransferase (ALT ) Serum Glutamic Pyruvate Transaminase (SGPT) ≤ 2.5 x upper limit of normal range (ULN); if hepatic metastases present ≤ 5.0 x ULN
    * Total serum bilirubin ≤ ULN; or total bilirubin ≤ 3.0 × ULN with direct bilirubin within normal range in subjects with documented Gilbert's Syndrome
    * Creatinine clearance > 60 mL/min (by Cockcroft-Gault)
15. Females of child-bearing potential [defined as a sexually mature women who (1) have not undergone hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or (2) have not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time during the preceding 24 consecutive months)] must:

    * Demonstrate a negative serum pregnancy test result at screening (performed by central lab) confirmed by local negative urine pregnancy dipstick within 72 hours prior to the first dose of IP); pregnancy test with sensitivity of at least 25 mIU/mL; and
    * Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis) or agree to use, and be able to comply with, two physician approved effective contraception methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) without interruption for 28 days or longer as required by local guidelines, prior to starting study drug, during the study therapy (including dose interruptions), and for 28 days after discontinuation of the study or longer as required by local guidelines
16. Females must abstain from breastfeeding starting at randomization, during study participation and for 28 days or longer as required by local guidelines, after IP discontinuation
17. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted
18. Able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. Male subjects
2. Concurrent chemotherapy or any other anti tumor therapy for breast cancer. Prior immunotherapy & monoclonal antibody therapy are acceptable.
3. Subjects who received prior cytotoxic chemotherapy after incomplete resection of locoregional recurrent disease
4. History of, or known current evidence of brain metastasis, including leptomeningeal involvement.
5. Subjects with bone as the only site of metastatic disease
6. Subjects with regional lymph node as the only site of metastatic disease
7. Serious intercurrent medical or psychiatric illness, including serious active infection
8. History of class II-IV congestive heart failure or myocardial infarction within 6 months of randomization
9. History of other primary malignancy in the last 5 years prior to randomization. Subjects with prior breast cancer history are eligible, however, the most recently obtained biopsy must demonstrate triple negative disease (source documented). Subjects with prior history of in situ cancer or basal or localized squamous cell skin cancer are eligible.
10. Subjects with a history of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple uncontrolled or unstable allergies which, in the opinion of the investigator, may lead to serious complications
11. Peripheral neuropathy Grade ≥ 2 by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0
12. Subjects who have received an investigational product within the previous 4 weeks prior to randomization
13. Subject is currently enrolled, or will enroll in a different clinical study in which investigational therapeutic procedures are performed or investigational therapies are administered while participating in this study
14. Pregnant or nursing women
15. Subjects with prior hypersensitivity to nab-paclitaxel, gemcitabine, carboplatin or any other platin, or nucleoside analogue agents
16. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
17. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if she were to participate in the study
18. Any condition that confounds the ability to interpret data from the study
19. History of seropositive human immunodeficiency virus (HIV)
20. Subjects who are receiving immunosuppressive or myelosuppressive medications that would, in the opinion of the investigator, increase the risk of serious neutropenic complications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2013-09-26 (Actual); Primary Completion 2016-10-28 (Actual); Study Completion 2016-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ileana Elias, M.D., Study Director — Celgene Corporation
Locations (140):
- United States (64):
  - Ironwood Cancer and Research Center, Chandler, Arizona
  - Arizona Center for Cancer Care, Glendale, Arizona
  - Arizona Cancer Research Alliance, Scottsdale, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Pacific Cancer Medical Center Inc, Anaheim, California
  - California Cancer Associates for Research and Excellence cCARE, Escondido, California
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Wilshire Oncology Medical Group, Inc, La Verne, California
  - Translational Research Management, Los Angeles, California
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Redwood Regional Medical Group, INC, Santa Rosa, California
  - Center for Hematology-Oncology, Boca Raton, Florida
  - Memorial Breast Cancer Center, Hollywood, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Joliet Oncology-Hematology Associates, Ltd, Joliet, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Investigative Clinical Research of Indiana, LLC, Indianapolis, Indiana
  - University of South Alabama Mitchell Cancer Institute, Lafayette, Louisiana
  - University of Maryland School of Med, Baltimore, Maryland
  - Center for Cancer and Blood Disorders, PC, Bethesda, Maryland
  - Henry Ford Medical Center - New Center One, Detroit, Michigan
  - Minnesota Oncology Hematology, PA, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Midwest Physicians Group, Kansas City, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - New Hampshire Oncology Hematology, Hooksett, New Hampshire
  - Dartmouth Hitchcock Medical Center Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hematology Oncology Associates of CNY, East Syracuse, New York
  - NYU Langone Arena Oncology, Lake Success, New York
  - Clinical Research Alliance, New York, New York
  - Alamance Regional Medical Cancer Center, Burlington, North Carolina
  - University of Cincinnatti, Cincinnati, Ohio
  - Oncology Hematology Care, Cincinnati, Ohio
  - Mark H Zangmeister Center, Columbus, Ohio
  - Toledo Community Oncology Program, Toledo, Ohio
  - Cancer Centers of Southwest Oklahoma, Lawton, Oklahoma
  - North Bend Medical Center, Coos Bay, Oregon
  - Northwest Cancer Specialists, P.C. - Hoyt, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - St Mary Medical Center, Langhorne, Pennsylvania
  - Magee Women's Hospital, Pittsburgh, Pennsylvania
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Texas Oncology, PA, Dallas, Texas
  - Texas Oncology, PA- Dallas, Dallas, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - UT Physicians General Medicine, Houston, Texas
  - Cancer Care Centers of South Texas - Loop, San Antonio, Texas
  - Texas Oncology P.A.- Tyler, Tyler, Texas
  - Hematology Oncology Associates of Fredericksburg, Fredericksburg, Virginia
  - Delta Hematologyoncology Associates, Portsmouth, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Medical Oncology Associates, Spokane, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Columbia St Marys Cancer Center, Milwaukee, Wisconsin
- Australia (4):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Frankston Hospital Oncology Research, Frankston, Victoria
  - Border Medical Oncology, Wodonga, Victoria
  - Sir Charles Gairdner Hospital, Nedlands
- Austria (3):
  - Universitaetsklinik Innsbruck, Innsbruck
  - Salzburger Landkliniken St. Johanns-Spital, Salzburg
  - Medizinische Universitat Wien, Vienna
- Brazil (15):
  - Centro de Oncologia Da Bahia, Salvador, Estado de Bahia
  - Liga Paranaense de Combate Ao Cancer, Curitiba, Paraná
  - Instituto Nacional de Cancer - INCA, Rio de Janerio, Rio de Janeiro
  - Associacao Hospitalar Moinhos de Vento Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Hospital Dr. Amaral Carvalho/ Hospital Amaral Carvalho Jaú, Jau/SP, São Paulo
  - ONCOCLINIC Clinica de Oncologia LTDA, Fortaleza
  - Instituto Ribeiraopretano de Combate Ao Cancer, Ribeirão Preto
  - Hospital das Clinicas da Faculdade de Medicina da USP, Ribeirão Preto
  - Hospital Bruno Born, Rio Grande
  - Hospital de Base Da Faculdade de Medicina de, São José do Rio Preto
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo
  - Instituto Brasileiro de Controle Do Cancer IBCC, São Paulo
  - Hospital Albert Einstein Sociedade Beneficente Israelita Brasileira, São Paulo
- Canada (5):
  - Ottawa General Hospital, Ottawa, Ontario
  - CHUM - Notre Dame, Montreal, Quebec
  - Hospital du Saint Scarement Sacrement Laboratory, Québec, Quebec
  - CSSS de Rimouski Neigette, Rimouski, Quebec
  - Alan Blair Cancer Centre at Pasqua Hosptial, Regina, Saskatchewan
- Centre Jean Perrin, Clermont-Ferrand, France
- Germany (10):
  - Sankt Gertrauden-Krankenhaus, Berlin
  - Facharztpraxis fur Gynakologie und Geburtshilfe, Bonn
  - Schwerpunktpraxis fur Gynakologische Onkologie, Cologne
  - Agaplesion Markus Krankenhaus, Frankfurt
  - Praxis fur interdisziplinare Onkologie & Hamatologie, Freiburg im Breisgau
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Frauenarzte am Bahnhofsplatz, Hildesheim
  - LMU Klinikum der Universitat, München
  - Krankenanstalt Mutterhaus der Borromaerinnen, Trier
  - Universitatsklinikum Ulm, Ulm
- Greece (5):
  - University of Athens Medical school - Regional General Hospital, Athens
  - IASO General, Athens
  - Metropolitan Hospital, Faliro
  - University General Hospital of Heraklion, Heraklion
  - University General Hospital of Patras, Rio Patras
- Italy (16):
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico S.Orsola-Malpighi, Bologna, Emilia-Romagna
  - Azienda Ospedaliero-Universitaria di Ferrara Arcispedale Sant' Anna, Ferrara
  - IRCCS AziendaOspedaliera Universitaria San Martino, Genova
  - Presidio Ospedaliero della Misericordia, Grosseto
  - Azienda Ospedaliera Ospedali Riuniti Papardo-Piemonte, Messina
  - Azienda Ospedaliera San Gerardo, Monza
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - Istituto Nazionale Per Lo Studio E La Cura Dei Tumori Fondazione Giovanni Pascale, Napoli, Campania
  - Istituto Oncologico Veneto, Padua
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Policlinico Universitario A Gemelli, Roma
  - Azienda Ospedaliera Sant Andrea, Roma
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Istituto Clinico Humanitas, Rozzano (MI)
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino, Torino, Piemonte
  - Azienda Ospedaliera Treviglio-Caravaggio, Treviglio
- Portugal (4):
  - Hospital Espirito Santo, Evora
  - Hospital Da Luz, Lisbon
  - Hospital de Santa Maria, Lisbon
  - Instituto Portugues de Oncologia do Porto, Francisco Gentil, Porto
- Spain (8):
  - Clinic Barcelona Hospital Universitari, Barcelona
  - Hospital Universitario Vall D Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Onkologikoa - Kutxaren Institutu Onkologikoa, Donostia / San Sebastian
  - Hospital General Gregorio Maranon, Madrid
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (5):
  - Royal United Hospital, Bath
  - Sarah Cannon Research Institute UK, London
  - The Christie NHS Foundation Trust, Manchester
  - The East and North Hertfordshire NHS Trust, Middlesex
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield South Yorkshire

REFERENCES:
- [Background] Yardley DA, Brufsky A, Coleman RE, Conte PF, Cortes J, Gluck S, Nabholtz JM, O'Shaughnessy J, Beck RM, Ko A, Renschler MF, Barton D, Harbeck N. Phase II/III weekly nab-paclitaxel plus gemcitabine or carboplatin versus gemcitabine/carboplatin as first-line treatment of patients with metastatic triple-negative breast cancer (the tnAcity study): study protocol for a randomized controlled trial. Trials. 2015 Dec 16;16:575. doi: 10.1186/s13063-015-1101-7. PMID 26673577
- [Derived] Liu MC, Janni W, Georgoulias V, Yardley DA, Harbeck N, Wei X, McGovern D, Beck R. First-Line Doublet Chemotherapy for Metastatic Triple-Negative Breast Cancer: Circulating Tumor Cell Analysis of the tnAcity Trial. Cancer Manag Res. 2019 Dec 12;11:10427-10433. doi: 10.2147/CMAR.S208712. eCollection 2019. PMID 31849532

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted by investigators in 11 countries in North America, Europe, Australia and South America, and enrolled participants at a total of 86 sites.
  Due to changes in the treatment landscape since the initiation of this trial, the decision was made not to proceed to the Phase 3 portion of the study.
Pre-assignment Details: Participants were randomized 1:1:1, stratified by disease free interval (≤ 1 year; > 1 year).
Groups:
- Arm A: Nab-Paclitaxel Plus (+) Gemcitabine: Participants received nab-Paclitaxel 125 mg/m^2 on Days 1 and 8 by intravenous (IV) administration followed by gemcitabine 1000 mg/m^2 on Days 1 and 8 by IV administration in each 21-day treatment cycle. Participants continued treatment until progressive disease (PD), unacceptable toxicity, required palliative radiotherapy or surgical intervention of lesion(s), withdrawal from study treatment, withdrawal of study consent, participant refusal or the investigator felt it was no longer in the best interest of the participant to continue on treatment.
- Arm B: Nab-Paclitaxel + Carboplatin: Participants received nab-Paclitaxel 125 mg/m^2 on Days 1 and 8 by IV administration followed by carboplatin area under the curve 2 (AUC 2) on Days 1 and 8 in each 21-day treatment cycle. Participants continued treatment until progressive disease (PD), unacceptable toxicity, required palliative radiotherapy or surgical intervention of lesion(s), withdrawal from study treatment, withdrawal of study consent, participant refusal or the investigator felt it was no longer in the best interest of the participant to continue on treatment.
- Arm C: Gemcitabine + Carboplatin: Participants received gemcitabine 1000 mg/m^2 on Days 1 and 8 by IV administration, followed by carboplatin AUC 2 on Days 1 and 8 by IV administration in each 21-day treatment cycle. Participants continued treatment until progressive disease (PD), unacceptable toxicity, required palliative radiotherapy or surgical intervention of lesion(s), withdrawal from study treatment, withdrawal of study consent, participant refusal or the investigator felt it was no longer in the best interest of the participant to continue on treatment.
Period: Overall Study
Arm/Group | Arm A: Nab-Paclitaxel Plus (+) Gemcitabine | Arm B: Nab-Paclitaxel + Carboplatin | Arm C: Gemcitabine + Carboplatin
Started | 61 | 64 | 66
Safety Population | 60 (Safety Population = randomized who received at least 1 dose of Investigational Product (IP)) | 64 (Safety Population = randomized who received at least 1 dose of IP) | 64 (Safety Population = randomized who received at least 1 dose of IP)
Treatment Discontinued | 60 (Treatment Duration=PD, toxicity, radiation/removal of lesions, consent withdrawal, doctor decision) | 64 (Treatment Duration=PD, toxicity, radiation/removal of lesions, consent withdrawal, doctor decision) | 64 (Treatment Duration=PD, toxicity, radiation/removal of lesions, consent withdrawal, doctor decision)
Completed | 0 (Not applicable according to the study design) | 0 (Not applicable according to the study design) | 0 (Not applicable according to the study design)
Not Completed | 61 | 64 | 66
Not completed — Death | 2 | 0 | 1
Not completed — Adverse Event | 9 | 13 | 12
Not completed — Progressive Disease | 31 | 35 | 36
Not completed — Symptomatic Deterioration | 3 | 3 | 1
Not completed — Withdrawal by Subject | 6 | 4 | 6
Not completed — Physician Decision | 4 | 3 | 6
Not completed — Non-Compliance with Study Drug | 1 | 2 | 0
Not completed — Given Commercially Available Drug | 0 | 0 | 2
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Miscellaneous | 3 | 3 | 0
Not completed — Untreated: Other | 0 | 0 | 1
Not completed — Untreated: Death | 0 | 0 | 1
Not completed — Untreated: Withdrawal Before Study Start | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population includes all randomized participants regardless of whether they received any IP or had any efficacy assessments collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Nab-Paclitaxel Plus (+) Gemcitabine | Arm B: Nab-Paclitaxel + Carboplatin | Arm C: Gemcitabine + Carboplatin | Total
Number analyzed (Participants) | 61 | 64 | 66 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (12.16) | 54.3 (11.96) | 56.7 (10.87) | 54.9 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 64 | 66 | 191
  Male | 0 | 0 | 0 | 0
Race [Count of Participants; unit: Participants]
  Black or African American | 9 | 6 | 8 | 23
  White | 50 | 55 | 54 | 159
  Unknown or Not Reported | 2 | 3 | 4 | 9
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status is used by doctors and researchers to assess how a subject's disease is progressing, assess how the disease affects the daily living activities of the subject and determine appropriate treatment and prognosis. 0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care (Least Favorable Activity)
  Participants
    0 = Fully Active | 34 | 38 | 42 | 114
    1 = Restrictive but ambulatory | 25 | 26 | 22 | 73
    2 = Ambulatory but unable to work | 1 | 0 | 0 | 1
    Missing | 1 | 0 | 2 | 3
Disease Free Interval by Clinical Interpretation [Number; unit: Years] — Disease Free Interval is defined as period of being absent of disease less than or equal to one year or free of disease greater than one year.
  Years
    ≤ 1 year | 17 | 16 | 20 | 53
    > 1 year | 43 | 48 | 45 | 136
    Missing | 1 | 0 | 1 | 2
Time from Diagnosis to First Documented Disease/Relapse [Mean (Standard Deviation); unit: months] | 38.8 (49.46) | 29.9 (37.18) | 50.9 (62.60) | 40.0 (51.46)
Time from First Documented Metastatic Disease/Relapse to Study Randomization [Mean (Standard Deviation); unit: months] | 2.1 (5.08) | 4.2 (18.39) | 1.6 (1.70) | 2.6 (11.07)
Time from Primary Diagnosis to Randomization [Mean (Standard Deviation); unit: months] | 43.7 (54.60) | 35.5 (40.51) | 52.5 (62.37) | 44.0 (53.53)
Current Sites of Metastasis [Number; unit: participants]
  Lymph Nodes(s) | 38 | 50 | 51 | 139
  Lung/Thoracic | 42 | 42 | 41 | 125
  Bone | 23 | 21 | 25 | 69
  Liver | 17 | 16 | 23 | 56
  Right/Left Breast | 15 | 19 | 17 | 51
  Skin/Soft Tissue | 13 | 13 | 8 | 34
  Other | 13 | 10 | 8 | 31
  Abdomen/Peritoneal | 1 | 2 | 3 | 6
Stage of Primary Diagnosis [Count of Participants; unit: Participants] — Invasive breast cancer stages:
  * Stage 0-Stage 0 = noninvasive ductal carcinoma in situ
  * Stage Ia-cancer cells are breaking through to or invading normal surrounding breast tissue.
  * Stage IIa-breast tumor about 2cm and involvement of ancillary lymph nodes.
  * Stage IIb-a larger tumor than earlier phases.
  * Stage IIIa-axillary lymph nodes clumping together.
  * Stage IIIb-spread further to the skin, breast bone or chest wall.
  * Stage IIIc-expanded involvement of lymph nodes.
  * Stage IV-cancer that has spread beyond the breast and nearby lymph nodes to other organs of the body.
  Participants
    Stage 0 | 0 | 1 | 0 | 1
    Stage IA | 7 | 6 | 11 | 24
    Stage IB | 0 | 0 | 0 | 0
    Stage IIA | 14 | 9 | 15 | 38
    Stage IIB | 8 | 7 | 9 | 24
    Stage IIIA | 9 | 10 | 3 | 22
    Stage IIIB | 3 | 3 | 5 | 11
    Stage IIIC | 3 | 3 | 2 | 8
    Stage IV | 11 | 17 | 10 | 38
Triple-Negative Breast Cancer (TNBC) at Primary Diagnosis [Count of Participants; unit: Participants] — Triple-Negative Breast Cancer defined as estrogen receptor (ER) negative, progesterone receptor (PgR) negative, and human epidermal growth factor receptor 2 (HER2) negative.
  Participants | 51 | 53 | 48 | 152
Triple-Negative at Latest Diagnosis [Count of Participants; unit: Participants] | 60 | 62 | 65 | 187

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimates of Progression-Free Survival (PFS) Based on Investigator Assessment.
Description: PFS was defined as the time from the date of randomization to the date of disease progression or death from any cause on or prior to the data cutoff date for the statistical analysis, whichever occurred earlier. Tumor responses were assessed every 6 weeks using, Response Evaluation Criteria in Solid Tumors (RECIST 1.1) and defined as: Complete response (CR) is the disappearance of all target lesions; Partial response (PR) occurs when at least a 30% decrease in the sum of diameters of target lesions from baseline; Stable disease is neither sufficient shrinkage to qualify for a PR nor sufficient increase of lesions to qualify for Progressive disease (PD); Progressive Disease- is at least a 20% increase in the sum of diameters of target lesions from nadir.
Time Frame: From date of randomization to data cut-off date of 16 December 2016; total length of time on study was 31 months for Arm A, 34 months for Arm B and 35 months for Arm C
Population: ITT includes all randomized participants regardless of whether they received any IP or had any efficacy assessments collected. Those who did not have disease progression or had not died as of the data cutoff date were censored at the time of the last radiologic assessment prior to the data cutoff date.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm A: Nab-Paclitaxel + Gemcitabine: Participants received nab-Paclitaxel 125 mg/m^2 on Days 1 and 8 by intravenous (IV) administration followed by gemcitabine 1000 mg/m^2 on Days 1 and 8 by IV administration of each 21-day treatment cycle. Participants continued treatment until progressive disease (PD), unacceptable toxicity, required palliative radiotherapy or surgical intervention of lesion(s), withdrawal from study treatment, withdrawal of study consent, participant refusal or the investigator felt it was no longer in the best interest of the participant to continue on treatment
Arm/Group | Arm A: Nab-Paclitaxel + Gemcitabine | Arm B: Nab-Paclitaxel + Carboplatin | Arm C: Gemcitabine + Carboplatin
Number analyzed (Participants) | 61 | 64 | 66
months | 5.5 [4.1 to 7.0] | 8.3 [5.7 to 10.6] | 6.0 [4.7 to 7.2]
Statistical Analysis 1: Comparison: Arm A: Nab-Paclitaxel + Gemcitabine vs Arm B: Nab-Paclitaxel + Carboplatin; For stratified analysis, the stratified log-rank test and stratified Cox proportional hazards model were used, where the stratification factor is the disease free interval (<= 1 year; > 1 year); Test type: Superiority or Other; p = 0.0183, Log Rank; Hazard Ratio (HR) = 1.692, 95% CI 2-sided [1.089 to 2.629]
Statistical Analysis 2: Comparison: Arm B: Nab-Paclitaxel + Carboplatin vs Arm C: Gemcitabine + Carboplatin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0152, Log Rank; Hazard Ratio (HR) = 0.581, 95% CI 2-sided [0.373 to 0.904]
Statistical Analysis 3: Comparison: Arm A: Nab-Paclitaxel + Gemcitabine vs Arm C: Gemcitabine + Carboplatin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8599, Log Rank; Hazard Ratio (HR) = 1.039, 95% CI 2-sided [0.676 to 1.597]

2. Secondary Outcome: Percentage of Participants With an Objective Complete or Partial Overall Response by Investigator Assessment.
Description: Percentage of participants with an Objective Complete or Partial Overall Response according to RECIST 1.1 and defined as: Complete response-disappearance of all target lesions; partial response at least a 30% decrease in the sum of diameters of target lesions from baseline; stable disease-neither sufficient shrinkage to qualify for PR nor sufficient increase of lesions to qualify for Progressive disease (PD)• Progressive Disease- At least a 20% increase in the sum of diameters of target lesions from nadir.
Time Frame: Disease response was assessed every 6 weeks; from date of randomization to data cut-off date of 16 December 2016; total length of time on study was 31 months for Arm A, 34 months for Arm B and 35 months for Arm C
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Nab-Paclitaxel + Gemcitabine | Arm B: Nab-Paclitaxel + Carboplatin | Arm C: Gemcitabine + Carboplatin
Number analyzed (Participants) | 61 | 64 | 66
percentage of participants | 39.3 [27.1 to 52.7] | 73.4 [60.9 to 83.7] | 43.9 [31.7 to 56.7]

3. Secondary Outcome: Percentage of Participants Who Initiated Cycle 6 Receiving Doublet Combination Therapy
Description: The percentage of participants who initiated Cycle 6 receiving doublet combination therapy regardless of the need for dose modifications.
Time Frame: Cycle 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Nab-Paclitaxel + Gemcitabine | Arm B: Nab-Paclitaxel + Carboplatin | Arm C: Gemcitabine + Carboplatin
Number analyzed (Participants) | 61 | 64 | 66
percentage of participants | 55.7 [42.5 to 68.5] | 64.1 [51.1 to 75.7] | 50.0 [37.4 to 62.6]

4. Secondary Outcome: Kaplan-Meier Estimates of Overall Survival
Description: Overall survival was defined as the time from the date of randomization to the date of death (from any cause).
Time Frame: as for outcome 1
Population: The ITT population includes all randomized participants regardless of whether the participant received any Investigational Product (IP) or had any efficacy assessments collected.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Nab-Paclitaxel + Gemcitabine | Arm B: Nab-Paclitaxel + Carboplatin | Arm C: Gemcitabine + Carboplatin
Number analyzed (Participants) | 61 | 64 | 66
months | 12.1 [9.4 to 15.9] | 16.8 [11.3 to 20.6] | 12.6 [10.1 to 16.6]
Statistical Analysis 1: Comparison: Arm A: Nab-Paclitaxel + Gemcitabine vs Arm B: Nab-Paclitaxel + Carboplatin; Hazard ratios and associated two-sided 95% confidence intervals were estimated using stratified Cox proportional hazard model. The stratification factor is the disease free interval (≤ 1 year; > 1 year); Test type: Superiority or Other; p = 0.1579, Log Rank; Hazard Ratio (HR) = 1.375, 95% CI 2-sided [0.882 to 2.143]
Statistical Analysis 2: Comparison: Arm B: Nab-Paclitaxel + Carboplatin vs Arm C: Gemcitabine + Carboplatin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.2945, Log Rank; Hazard Ratio (HR) = 0.796, 95% CI 2-sided [0.520 to 1.221]
Statistical Analysis 3: Comparison: Arm A: Nab-Paclitaxel + Gemcitabine vs Arm C: Gemcitabine + Carboplatin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.6691, Log Rank; Hazard Ratio (HR) = 1.101, 95% CI 2-sided [0.710 to 1.708]

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Treatment-emergent adverse events (TEAEs) were defined as any AEs that began or worsened with the onset date on or after the date of the first dose of IP through 28 days after the last dose. A serious AE (SAE) = any AE which results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event. The severity of AEs was graded based on the participant's symptoms according to the Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0); AEs were evaluated for severity as follows: Grade 1 = Mild - transient or mild discomfort; no medical intervention required; Grade 2 = Moderate - mild to moderate limitation in activity; Grade 3 = Severe; Grade 4 = Life threatening; Grade 5 = Death.
Time Frame: From randomization through to 28 days after the last dose of IP; up to data cut off date of 16 Dec 2016; maximum treatment duration of study drug exposure was 108.3 weeks for Arm A, 83 weeks for Arm B, 110.1 weeks for Arm C
Population: The safety population includes all randomized participants who received at least 1 dose of IP.
Measure: Number; unit: participants
Arm/Group | Arm A: Nab-Paclitaxel + Gemcitabine | Arm B: Nab-Paclitaxel + Carboplatin | Arm C: Gemcitabine + Carboplatin
Number analyzed (Participants) | 60 | 64 | 64
participants
  Any TEAE | 60 | 63 | 64
  Any Grade 3 or Higher TEAE | 46 | 51 | 54
  Treatment-related TEAE | 59 | 62 | 60
  Treatment-related, Grade 3 or Higher TEAE | 35 | 43 | 46
  Serious TEAE | 22 | 20 | 25
  Treatment-related Serious TEAE | 10 | 9 | 13
  TEAE Leading to Discontinuation (D/C) of IP | 16 | 29 | 15
  Treatment Related (TR) TEAE Leading to D/C of IP | 12 | 27 | 12
  TEAE Leading to Dose Reduction (DR) of IP | 23 | 20 | 25
  Treatment related TEAE Leading to DR of IP | 23 | 20 | 23
  TEAE Leading to Dose Interruption (DI) of IP | 31 | 50 | 50
  TR TEAE Leading to DI of IP | 27 | 44 | 44
  TEAE leading to D/C of nab-Paclitaxel | 16 | 17 | 0
  TR TEAE leading to D/C of nab-Paclitaxel | 11 | 13 | 0
  TEAE leading to DR of nab-Paclitaxel | 22 | 19 | 0
  TR TEAE leading to DR of nab-Paclitaxel | 21 | 19 | 0
  TEAE leading to DI of nab-Paclitaxel | 31 | 50 | 0
  TR TEAE leading to DI of nab-Paclitaxel | 27 | 44 | 0
  TEAE leading to D/C of Gemcitabine | 13 | 0 | 13
  TR TEAE leading to D/C of Gemcitabine | 7 | 0 | 9
  TEAE leading to DR of Gemcitabine | 18 | 0 | 25
  TR TEAE leading to DR of Gemcitabine | 18 | 0 | 23
  TEAE leading to DI of Gemcitabine | 31 | 0 | 49
  TR TEAE leading to DI of Gemcitabine | 24 | 0 | 43
  TEAE leading to D/C of Carboplatin | 0 | 28 | 15
  TR TEAE leading to D/C of Carboplatin | 0 | 25 | 12
  TEAE leading to DR of Carboplatin | 0 | 17 | 21
  TR TEAE leading to DR of Carboplatin | 0 | 17 | 20
  TEAE leading to DI of Carboplatin | 0 | 50 | 50
  TR TEAE leading to DI of Carboplatin | 0 | 44 | 43
  TEAE Leading to Death | 2 | 1 | 2
  Treatment Related TEAE leading to death | 1 | 0 | 1

6. Secondary Outcome: Percentage of Participants Experiencing Dose Modifications (Reductions and Interruptions)
Description: The number of participants with dose modifications occurring during the treatment period. Dose reductions and interruptions are typically caused by clinically significant laboratory abnormalities and /or treatment emergent adverse events/toxicities.
Time Frame: From randomization through to 28 days after the last dose of IP; up to data-cut off of date of 16 Dec 2016; maximum treatment duration of study drug exposure was 108.3 weeks for Arm A, 83 weeks for Arm B, 110.1 weeks for Arm C
Population: The Safety/Treated population includes all randomized participants who received at least 1 dose of IP.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Nab-Paclitaxel + Gemcitabine | Arm B: Nab-Paclitaxel + Carboplatin | Arm C: Gemcitabine + Carboplatin
Number analyzed (Participants) | 60 | 64 | 64
percentage of participants
  ≥ one DR for both IPs | 33.3 | 46.9 | 51.6
  ≥ one DI for both IPs | 38.3 | 70.3 | 73.4
  ≥ one dose missed for both IPs | 48.3 | 45.3 | 56.3

7. Secondary Outcome: Percentage of Participants Who Discontinued From All Study Treatment Due to TEAEs
Description: Treatment-emergent adverse events (TEAEs) were defined as any AEs that begin or worsen with an onset date on or after the date of the first dose of IP through 28 days after the last dose.
Time Frame: as for outcome 6
Population: The Safety/Treated population includes all randomized participants who received at least 1 dose of IP.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Nab-Paclitaxel + Gemcitabine | Arm B: Nab-Paclitaxel + Carboplatin | Arm C: Gemcitabine + Carboplatin
Number analyzed (Participants) | 60 | 64 | 64
percentage of participants | 21.7 [12.1 to 34.2] | 26.6 [16.3 to 39.1] | 21.9 [12.5 to 34.0]

ADVERSE EVENTS:
Time Frame: From randomization through to 28 days after the last dose of IP; up to the data cut-off date of 16 December 2016; AEs collected and monitored for 39 months.
Description: Maximum treatment duration of study drug exposure was 108.3 weeks for Arm A, 83 weeks for Arm B and 110.1 weeks for Arm C
Groups:
- Arm A: Nab-Paclitaxel + Gemcitabine: Participants received nab-Paclitaxel 125 mg/m^2 on Days 1 and 8 by intravenous (IV) administration followed by gemcitabine 1000 mg/m^2 on Days 1 and 8 by IV administration in each 21-day treatment cycle.
- Arm B: Nab-Paclitaxel + Carboplatin: Participants received nab-Paclitaxel 125 mg/m^2 on Days 1 and 8 by IV administration followed by Carboplatin AUC 2 on Days 1 and 8 in each 21-day treatment cycle.
- Arm C: Gemcitabine + Carboplatin: Participants received Gemcitabine 1000 mg/m^2 on Days 1 and 8 by IV administration, followed by carboplatin AUC 2 on Days 1 and 8 by IV administration in each 21-day treatment cycle.
Arm/Group | Arm A: Nab-Paclitaxel + Gemcitabine | Arm B: Nab-Paclitaxel + Carboplatin | Arm C: Gemcitabine + Carboplatin
Serious Adverse Events (participants affected / at risk) | 22/60 | 20/64 | 25/64
Other Adverse Events (participants affected / at risk) | 59/60 | 63/64 | 62/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nab-Paclitaxel + Gemcitabine (N=60) | Arm B: Nab-Paclitaxel + Carboplatin (N=64) | Arm C: Gemcitabine + Carboplatin (N=64)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Fatigue (General disorders) | 1 | 0 | 1
General physical health deterioration (General disorders) | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 2
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 4 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Nodular regenerative hyperplasia (Hepatobiliary disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Breast cellulitis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 1 | 0 | 0
Device related sepsis (Infections and infestations) | 1 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 4 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Sepsis (Infections and infestations) | 1 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Sensory disturbance (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nab-Paclitaxel + Gemcitabine (N=60) | Arm B: Nab-Paclitaxel + Carboplatin (N=64) | Arm C: Gemcitabine + Carboplatin (N=64)
Anaemia (Blood and lymphatic system disorders) | 25 | 33 | 30
Leukopenia (Blood and lymphatic system disorders) | 4 | 12 | 14
Lymphopenia (Blood and lymphatic system disorders) | 1 | 6 | 5
Neutropenia (Blood and lymphatic system disorders) | 24 | 43 | 44
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 18 | 34
Tachycardia (Cardiac disorders) | 3 | 1 | 3
Lacrimation increased (Eye disorders) | 1 | 4 | 1
Vision blurred (Eye disorders) | 3 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 9 | 5
Abdominal pain upper (Gastrointestinal disorders) | 5 | 7 | 5
Constipation (Gastrointestinal disorders) | 13 | 27 | 25
Diarrhoea (Gastrointestinal disorders) | 25 | 26 | 13
Dry mouth (Gastrointestinal disorders) | 3 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 2 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 1 | 1
Nausea (Gastrointestinal disorders) | 26 | 34 | 27
Stomatitis (Gastrointestinal disorders) | 5 | 14 | 8
Vomiting (Gastrointestinal disorders) | 18 | 13 | 11
Asthenia (General disorders) | 13 | 10 | 15
Chills (General disorders) | 4 | 3 | 2
Fatigue (General disorders) | 33 | 32 | 24
Generalised oedema (General disorders) | 3 | 0 | 0
Influenza like illness (General disorders) | 3 | 4 | 2
Non-cardiac chest pain (General disorders) | 6 | 3 | 2
Oedema peripheral (General disorders) | 17 | 12 | 10
Pain (General disorders) | 3 | 3 | 6
Pyrexia (General disorders) | 12 | 5 | 8
Drug hypersensitivity (Immune system disorders) | 3 | 9 | 2
Hypersensitivity (Immune system disorders) | 0 | 5 | 0
Bronchitis (Infections and infestations) | 2 | 5 | 1
Cellulitis (Infections and infestations) | 4 | 2 | 0
Folliculitis (Infections and infestations) | 4 | 1 | 0
Influenza (Infections and infestations) | 1 | 4 | 2
Sinusitis (Infections and infestations) | 3 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 7 | 2
Urinary tract infection (Infections and infestations) | 3 | 11 | 6
Contusion (Injury, poisoning and procedural complications) | 1 | 5 | 1
Fall (Injury, poisoning and procedural complications) | 4 | 5 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 6 | 2
Alanine aminotransferase increased (Investigations) | 6 | 0 | 5
Aspartate aminotransferase increased (Investigations) | 6 | 0 | 4
Weight decreased (Investigations) | 8 | 4 | 3
Decreased appetite (Metabolism and nutrition disorders) | 15 | 14 | 10
Dehydration (Metabolism and nutrition disorders) | 6 | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 5 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 12 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 12 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 9 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 14 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 5 | 8
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 14 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 7 | 4
Spinal pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 11 | 9
Dysgeusia (Nervous system disorders) | 9 | 9 | 4
Headache (Nervous system disorders) | 17 | 14 | 12
Hypoaesthesia (Nervous system disorders) | 2 | 4 | 2
Neuropathy peripheral (Nervous system disorders) | 4 | 11 | 3
Neurotoxicity (Nervous system disorders) | 4 | 3 | 0
Paraesthesia (Nervous system disorders) | 4 | 7 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 14 | 14 | 5
Anxiety (Psychiatric disorders) | 3 | 2 | 3
Depression (Psychiatric disorders) | 4 | 2 | 7
Insomnia (Psychiatric disorders) | 8 | 12 | 11
Breast pain (Reproductive system and breast disorders) | 0 | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 17 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 15 | 11
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 33 | 25 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 4 | 5 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 9 | 4
Rash (Skin and subcutaneous tissue disorders) | 8 | 3 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 4
Hot flush (Vascular disorders) | 4 | 5 | 2
Hypertension (Vascular disorders) | 8 | 4 | 1
Lymphoedema (Vascular disorders) | 2 | 6 | 3

LIMITATIONS AND CAVEATS:
Due to changes in the treatment landscape since the trial initiation, including the initiation of trials with immunotherapy drugs, successful enrollment of the Phase 3 part was considered unlikely and was not conducted; no safety signals were raised.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 12 months since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for 90 more days. Investigator must delete confidential information before submission or defer publication to permit patent applications.